CLINICAL TRIAL: NCT00857610
Title: Molecular Analyses of Retinoid-induced Dermatitis in Aged/Photoaged Human Skin
Brief Title: Retinol-induced Dermatitis in Aged Skin
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dana L. Sachs, MD, Professor of Dermatology, University of Michigan
Other Study IDs: HUM00026851/ Derm 604
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Aged Skin; Photoaged Skin
Keywords: Aged skin; Photoaged skin; Retinol; Topical retinoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies will be taken; however, they are not intended to be used for DNA extraction.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Subjects using 0.1% retinol one day per week
- 2: Subjects using 0.1% retinol three days per week
- 3: Subjects using 0.1% retinol seven days per week
- 4: Subjects using 0.5% retinol one day per week
- 5: Subjects using 0.5% retinol three days per week
- 6: Subjects using 0.5% retinol seven times per week

SUMMARY:
Topical therapy with retinoids is the only proven medical therapy for aged/photoaged human skin. However, topical therapy with retinoids often result in unwanted cutaneous dermatitis, including erythema and scaling. The reseachers intend to investigate the dose, frequency of use, and time dependence of topical retinol-induced dermatitis. The researchers intend to evaluate retinoid-induced dermatitis biochemically, including retinol regulation of retinoid responsive genes that control retinoid metabolism and serve as markers for retinoid bioactivity. The researchers will also investigate the role of EGF receptor pathway in retinoid-induced dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Subject is at least 21 years of age
* Good general health
* No disease states, physical conditions or medications that would impair evaluation of the test sites
* Willingness and ability to follow protocol
* Signed written and witnessed informed consent form
* No use of oral retnoids in the past year
* No use of topical steroids to the treatment area in the past 2 weeks

Exclusion Criteria:

* Has received an experimental drug or used and experimental device in the 14 days prior to admission to the study
* History of keloids
* History of hypersensitivity to lidocaine or epinephrine
* Pregnant or nursing women
* Disease states or physical condition that would impair evaluation of the test sites or compliance with the protocol
* History of chemical peels or laser treatments to the sites evaluated

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be between the ages of 21-60 years of age, with moderate clinical photodamage, and either gender.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2009-07-20 (Actual); Primary Completion 2014-08-29 (Actual); Study Completion 2014-08-29 (Actual)

PRIMARY OUTCOMES:
Retinoid-induced dermatitis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dana Sachs, MD, Principal Investigator — University of Michigan Professor of Dermatology
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States